CLINICAL TRIAL: NCT07191899
Title: Randomized, Single-blind, Placebo-controlled Exploratory Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety, Tolerability of KN060 in Patients With Essential Hypertension
Brief Title: To Evaluate the Efficacy and Safety of KN060 in Essential Hypertension
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KN060-D-102
Record Dates: First submitted 2025-06-06; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Essential hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.9% Sodium Chloride Injection (Placebo Comparator): 0.9% sodium chloride 100ml was administered as placebo by intravenous drip every two weeks
  Interventions: Drug: 0.9% Sodium Chloride Injection
- KN060 (Experimental): The dose was calculated based on the fasting body weight of the subject D1, and the corresponding volume of KN060 was drawn and added to 0.9% sodium chloride injection to prepare a 100 ml solution by intravenous drip every two weeks
  Interventions: Drug: KN060

INTERVENTIONS:
Drug: KN060 — The dose was calculated based on the fasting body weight of the subject D1, and the corresponding volume of KN060 was drawn and added to 0.9% sodium chloride injection to prepare a 100 ml solution by intravenous drip every two weeks
  Arms: KN060
Drug: 0.9% Sodium Chloride Injection — 0.9% sodium chloride 100ml was administered as placebo by intravenous drip every two weeks
  Arms: 0.9% Sodium Chloride Injection

SUMMARY:
The primary objective of this study is to compare the change from baseline in systolic blood pressure between KN060 and placebo in patients with essential hypertension over 12 weeks; the secondary objectives are to assess the safety and tolerability of KN060 and to assess the pharmacokinetic and pharmacodynamic properties and immunogenicity of KN060 in patients with essential hypertension.

The main questions it aims to answer are:

* To verify the efficacy of KN060 in patients with essential hypertension
* Safety of KN060 in Subjects Treated for Essential Hypertension Researchers will compare KN060 to placebo (0.9% sodium chloride 100ml) to assess the antihypertensive effect of KN060.

Subjects will :

* Receive KN060 or placebo by intravenous drip every two weeks for 6 doses.
* AOBP, 24hABPM, HBPM,and safety were monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. men or women ≥ 18 years of age and ≤ 65 years of age;
2. patients with essential hypertension who are not receiving drug therapy or are receiving stable monotherapy (stable therapy: no change in antihypertensive drugs and doses within 30 days before screening);
3. AOBP mean sitting SBP ≥ 140 and < 180 mmHg (at least 5 minutes rest before measurement, 3 measurements averaged over at least 1 minute apart) and mean SBP ≥ 130 and ≤ 160 mmHg at 24 hours ABPM;

Exclusion Criteria:

1. secondary hypertension: kidney disease, endocrine disease, cardiovascular disease and moderate to severe obstructive sleep apnea without CPAP treatment;
2. Grade 3 hypertension (severe): mean AOBP sitting SBP ≥ 180 mmHg, and/or DBP ≥ 110 mmHg; mean ABPM SBP > 160 mmHg, and/or mean DBP ≥ 100 mmHg;
3. Patients with a history of hypertensive emergencies, or hypertensive sub-emergencies who have severe hypertension with headache, chest tightness, irritability, and epistaxis;
4. high risk of bleeding or abnormal relevant indicators;
5. long-term use of anticoagulants or antiplatelet drugs, including aspirin at any dose, due to treatment;
6. currently using, or within 30 days before dosing or expected to use any drug or other component known to affect blood pressure during the study;
7. Type 2 diabetes with substandard blood glucose control: fasting blood glucose > 7.8 mmol/L, or 2-hour postprandial blood glucose/random blood glucose > 10.0 mmol/L, or HbA1c > 7%;
8. any cardiovascular event within 6 months prior to screening
9. unstable heart disease, such as uncontrolled symptomatic arrhythmia, atrial fibrillation, heart failure NYHA ≥ III, severe left ventricular hypertrophy, or a history of valvular heart disease;
10. 12-lead ECG showed significant abnormal heart rate, arrhythmia or myocardial ischemia;
11. echocardiography revealed heart failure:LVEF< 50%; abnormal ventricular diastolic function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Systolic Blood Pressure (SBP) Change From Baseline in 24hABPM Adding KN060 or Placebo for 12 Weeks | KN060 or placebo for 12 weeks

SECONDARY OUTCOMES:
Proportion of subjects achieving target blood pressure control, incidence of adverse events, pharmacokinetic, pharmacodynamic and immunogenicity characteristics of KN060 in patients with essential hypertension | 12 weeks
  Change from Baseline in Mean Diastolic Blood Pressure (DBP) at 24hABPM Proportion of patients with reductions from baseline in mean nighttime/daytime SBP by ABPM Proportion of patients achieving blood pressure targets by ABPM (24-hour mean blood pressure < 130/80 mmHg, daytime mean blood pressure < 135/85 mmHg, nighttime mean blood pressure < 120/70 mmHg) Change from Baseline in AOBP Mean Sitting SBP, DBP Proportion of patients achieving sitting blood pressure targets for AOBP (< 140/90 mmHg, < 130/80 mmHg) Incidence of adverse events (TEAEs), serious adverse events (SAEs) and drug-related adverse events (TRAEs) in each group during the trial (treatment period and follow-up period) Pharmacokinetics and pharmacodynamics of KN060 in patients with essential hypertension Immunogenicity of KN060 in Patients with Essential Hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, Doctor, Principal Investigator — Ruijin Hospital; Ningru Zhang, Doctor, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University; Caie Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science & Technology; Zhijuan Li, Doctor, Principal Investigator — The First Affiliated Hospital of Henan University of Science & Technology; Siyu Guan, Doctor, Principal Investigator — Xiang Yang Central Hospital; Lipeng Li, Doctor, Principal Investigator — Luoyang third people's Hospital; Jidong Zhang, Doctor, Principal Investigator — The Second Hospital of Hebei Medical University; ZhiJun Huang, Doctor, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No